CLINICAL TRIAL: NCT05898984
Title: A Single Dose, Randomized, Open-label, 3-Way Cross-over Clinical Pharmacology Study, to Evaluate the Systemic Exposure of BDP, Beclomethasone 17-monoproprionate, Formoterol Fumarate, and Glycopyrronium Bromide, After Inhalation of the Fixed Combination BDP/FF/GB HFA pMDI (CHF 5993) at Two Different Strengths and of BDP Hydrofluoroalkane (HFA), in Healthy Volunteers.
Brief Title: Clinical Study to Evaluate the Safety, Tolerability and the Concentration of the BDP (Beclomethasone Dipropionate), Active Metabolite of BDP, FF( Formoterol Fumarate) and GB (Glycopyrronium Bromide), After Inhalation of CHF 5993 at Two Different Doses and QVAR®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Collaborators: SGS S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CLI-05993AB8-01
Record Dates: First submitted 2023-04-14; First posted 2023-06-12 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — alpha-ketoisovalerate dehydrogenase phosphatase

STUDY DESIGN:
Intervention Model Description: The doses will be administered to all subjects in a crossover design. The doses administered as a single dose for the Test product (T: CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI) and Reference product 1 (R1: CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI) in this study are equivalent to the TDD authorised for asthma and the maximum TDD authorized for Reference product 2 (R2: BDP HFA [QVAR REDIHALER®, BDP 80 μg]) in regular treatment of asthma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single dose of CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI (T) (Experimental): CHF 5993 BDP/FF/GB 200/6/12.5 µg via pressurized metered dose inhaler: 4 inhalations alternated with 4 inhalations of CHF 5993 placebo, corresponding to 8 inhalations in total and giving a total daily dose (TDD) of BDP/FF/GB: 800/24/50 µg.
  Interventions: Drug: Test product (T):CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI
- single dose of CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI (R1) (Active Comparator): CHF 5993 BDP/FF/GB 100/6/12.5 µg via pressurized metered dose inhaler: 4 inhalations alternated with 4 inhalations of CHF 5993 placebo, corresponding to 8 inhalations in total and giving a TDD of BDP/FF/GB: 400/24/50 µg.
  Interventions: Drug: Reference product 1 (R1): CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI
- Single dose of BDP HFA (QVAR REDIHALER®, BDP 80 μg) (R2) (Active Comparator): BDP HFA (QVAR REDIHALER®, BDP 80 μg): pressurised, breath-actuated, metered dose aerosol with a dose counter): 8 inhalations (TDD of BDP: 640 µg ex-actuator, 800 µg ex valve).
  Interventions: Drug: Reference product 2 (R2): BDP HFA (QVAR REDIHALER®, BDP 80 μg)

INTERVENTIONS:
Drug: Test product (T):CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI — CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI with HFA 134a propellant (fixed combination of BDP [200 μg], FF [6 μg] and GB [12.5 μg] via pMDI): 4 inhalations alternated with 4 inhalations of CHF 5993 placebo, corresponding to 8 inhalations in total and giving a total daily dose (TDD) of BDP/FF/GB: 800/24/50 µg.
  Reference product 1 (R1): CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI with HFA 134a propellant (fixed combination of BDP [100 μg], FF [6 μg] and GB [12.5 μg] via pMDI): 4 inhalations alternated with 4 inhalations of CHF 5993 placebo, corresponding to 8 inhalations in total and giving a TDD of BDP/FF/GB: 400/24/50 µg.
  Reference product 2 (R2): BDP HFA (QVAR REDIHALER®, BDP 80 μg): pressurised, breath-actuated, metered dose aerosol with a dose counter): 8 inhalations (TDD of BDP: 640 µg ex-actuator, 800 µg ex valve).
  Arms: single dose of CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI (T)
Drug: Reference product 1 (R1): CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI — with HFA 134a propellant (fixed combination of BDP [100 μg], FF [6 μg] and GB [12.5 μg] via pMDI): 4 inhalations alternated with 4 inhalations of CHF 5993 placebo, corresponding to 8 inhalations in total and giving a TDD of BDP/FF/GB: 400/24/50 µg
  Other Names: Trimbow Medium Strenght (MS)®
  Arms: single dose of CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI (R1)
Drug: Reference product 2 (R2): BDP HFA (QVAR REDIHALER®, BDP 80 μg) — pressurised, breath-actuated, metered dose aerosol with a dose counter): 8 inhalations (TDD of BDP: 640 µg ex-actuator, 800 µg ex valve).
  Other Names: QVAR REDIHALER®
  Arms: Single dose of BDP HFA (QVAR REDIHALER®, BDP 80 μg) (R2)

SUMMARY:
The study is being conducted to compare the pharmacokinetic (PK) of BDP (and its main active metabolite B17MP), FF, and GB between CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI and CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI (pressurized Metered Dose Inhaler), to assess the proportionality of systemic exposure to BDP and B17MP (17-Monoproprionate), and the systemic exposure to FF and GB with increasing doses of BDP.

The study includes a QVAR REDIHALER® arm too.

DETAILED DESCRIPTION:
The main purpose of this study is to evaluate the systemic exposure to B17MP, FF, and GB as the area under the concentration-time curve from zero to time 't' where t is the last quantifiable time point (AUC0-t) and maximum plasma concentration (Cmax) across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg).

The secondary purposes of the study are:

1. To evaluate the pharmacokinetic profile of BDP and additional pharmacokinetic parameters of B17MP, FF, and GB across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg);
2. To compare the exposure to BDP and B17MP between the high dose BDP/FF/GB (total daily dose [TDD]: 800/24/50 µg) and the highest US-approved dose of QVAR (TDD 800 µg).
3. generate additional safety and tolerability information of the two CHF 5993 pDMI strengths, after a single dose.

Participation in the study will last for a maximum of 70 days for each subject (starting from randomization).

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent ;
* 18-55 years of age;
* Ability to understand the study procedures, the risks involved and ability to be trained to correctly use the inhalers.
* Body mass index of 19.0 to 30.0 kg/m2 (extremes inclusive), and body weight ≥50.0 kg;
* Non- or ex-smokers who smoked <5 pack-years and stopped smoking >1 year prior to screening;
* Good physical and mental status, determined based on the medical history and a general clinical examination;
* Vital signs within normal limits at screening: diastolic blood pressure (DBP) 40 to 90 mmHg, systolic blood pressure (SBP) 90 to 140 mmHg
* 12-Lead digitised electrocardiogram (ECG) in triplicate considered as normal (40 ≤ heart rate [HR] ≤110 beats per minute, 120 milliseconds [ms] ≤ PR interval [PR] ≤220 ms [PR ≤120 ms without a delta wave may be acceptable], QRS interval [QRS] ≤120 ms, and Fridericia corrected QT interval [QTcF] ≤450 ms for males and QTcF ≤470 ms for females).
* Lung function measurements within normal limits at screening: forced expiratory volume in the first second (FEV1) equal to or more than 80% of predicted for the subject's normal value according to the Global Lung Function Initiative, European Respiratory Society Task Force Lung Function Reference Values and FEV1/forced vital capacity ratio >0.70.
* Female subjects of non-chid bearing potential or females of childbearing potential with a negative pregnancy test and acceptable contraceptive methods.

Exclusion Criteria:

* Participation in another clinical study with an investigational drug in the 30 days or five half-lives of that investigational drug (whichever is longer) preceding the administration of the study treatment; longer and more appropriate time could be considered by the Investigator based on the terminal half-life (t1/2) and/or long-term toxicity of the previous investigational drug;
* Clinically relevant and uncontrolled respiratory, cardiac, hepatic, gastrointestinal, renal, endocrine, metabolic, neurologic or psychiatric disorders that may interfere with successful completion of this protocol according to the Investigator's judgment;
* Subjects with history of breathing problems (i.e. history of asthma including childhood asthma);
* Positive urine test for cotinine.
* Intake of non-permitted concomitant medications in the predefined period prior to screening, or prior to randomisation or the subject is expected to take non-permitted concomitant medications during the study;
* Presence of any current infection, or previous infection that resolved less than 7 days prior to screening or prior to randomisation;
* Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation used in the study;
* Subjects with medical diagnosis of narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that in the opinion of the Investigator would prevent use of anticholinergics;
* For females only: pregnant or lactating women.
* Subjects receiving treatment with any drug known to have a well defined potential for hepatotoxicity.
* Subjects using e-cigarettes within 6 months before screening.

Other Inclusion/exclusion criteria as defined by the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — At least 28 subjects will be males and at least 28 subjects will be females, to ensure gender representation.
Enrollment: 69 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
systemic exposure ( area under the concentration time curve from zero to time) to beclomethasone 17 monopropionate (B17MP), FF and GB | From pre-dose to 24 hours post dose for BDP/B17MP and from pre-dose to 72hours post dose for FF and GB
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI:
  To evaluate the systemic exposure to beclomethasone 17 monopropionate (B17MP), FF and GB as area under the concentration time curve from zero to time 't' where t is the last quantifiable time point (AUC0-t) across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg).
systemic exposure (maximum plasma concentration (Cmax) ) to beclomethasone 17 monopropionate (B17MP), FF and GB | From pre-dose to 24 hours post dose for BDP/B17MP and from pre-dose to 72hours post dose for FF and GB
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI:
  To evaluate the systemic exposure to beclomethasone 17 monopropionate (B17MP), FF and GB as maximum plasma concentration (Cmax) across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg).

SECONDARY OUTCOMES:
Area under the concentration-time curve from zero to infinity (AUC0-∞) of B17MP, FF and GB across two different dose strengths of CHF 5993. | From pre-dose to 24 hours post dose for BDP/B17MP and from pre-dose to 72hours post dose for FF and GB
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI:
  To evaluate the area under the concentration-time curve from zero to infinity (AUC0-∞) of B17MP, FF and GB across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg);
Time to Cmax (t max) of B17MP, FF and GB across two different dose strengths of CHF 5993. | From pre-dose to 24 hours post dose for BDP/B17MP and from pre-dose to 72hours post dose for FF and GB
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI:
  To evaluate the Time to Cmax (t max) of B17MP, FF and GB across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg);
Time to t1/2 of B17MP, FF and GB across two different dose strengths of CHF 5993. | From pre-dose to 24 hours post dose for BDP/B17MP and from pre-dose to 72hours post dose for FF and GB
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI:
  To evaluate the Time to t1/2 of B17MP, FF and GB across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg);
Area under the concentration time curve from zero to time 't' where t is the last quantifiable time point (AUC0-t) of BDP across two different dose strengths of CHF 5993 | From pre-dose to 24 hours post dose for BDP/B17MP and from pre-dose to 72hours post dose for FF and GB
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI:
  To evaluate Area under the concentration time curve from zero to time 't' where t is the last quantifiable time point (AUC0-t) of B17MP, FF and GB across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg);
Time to Cmax (t max) of BDP across two different dose strengths of CHF 5993 | From pre-dose to 24 hours post dose for BDP/B17MP and from pre-dose to 72hours post dose for FF and GB
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI:
  To Time to Cmax (t max) of B17MP, FF and GB across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg);
t max of BDP across two different dose strengths of CHF 5993 | From pre-dose to 24 hours post dose for BDP/B17MP and from pre-dose to 72hours post dose for FF and GB
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. CHF 5993 BDP/FF/GB 100/6/12.5 µg pMDI:
  To evaluate the tmax of B17MP, FF and GB across two different dose strengths of CHF 5993 BDP/FF/GB (200/6/12.5 μg and 100/6/12.5 μg);
Area under the concentration time curve from zero to time 't' where t is the last quantifiable time point (AUC0-t) of BDP after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg) | From pre-dose to 24 hours post dose
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. BDP HFA (QVAR REDIHALER®, BDP 80 µg):
  To compare the systemic exposure to BDP as Area under the concentration time curve from zero to time 't' where t is the last quantifiable time point (AUC0-t) for B17MP after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg);
Area under the concentration time curve from zero to time 't' where t is the last quantifiable time point (AUC0-t) of B17MP after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg); | From pre-dose to 24 hours post dose
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. BDP HFA (QVAR REDIHALER®, BDP 80 µg):
  To compare the systemic exposure to B17MP as Area under the concentration time curve from zero to time 't' where t is the last quantifiable time point (AUC0-t) for B17MP after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg);
maximum plasma concentration (Cmax) of BDP after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg); | From pre-dose to 24 hours post dose
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. BDP HFA (QVAR REDIHALER®, BDP 80 µg):
  To compare the systemic exposure to BDP as maximum plasma concentration (Cmax) for B17MP after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg);
maximum plasma concentration (Cmax) of B17MPafter a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg); | From pre-dose to 24 hours post dose
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. BDP HFA (QVAR REDIHALER®, BDP 80 µg):
  To compare the systemic exposure to B17MP as maximum plasma concentration (Cmax) for B17MP after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg);
t max of BDP after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg); | From pre-dose to 24 hours post dose
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. BDP HFA (QVAR REDIHALER®, BDP 80 µg):
  To compare the systemic exposure to BDP as t max after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg);
t max of BDP of B17MPafter a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg); | From pre-dose to 24 hours post dose
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. BDP HFA (QVAR REDIHALER®, BDP 80 µg):
  To compare the systemic exposure to B17MP as t max after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg);
Area under the concentration-time curve from zero to infinity (AUC0-∞) of B17MPafter a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg); | From pre-dose to 24 hours post dose
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. BDP HFA (QVAR REDIHALER®, BDP 80 µg):
  To compare the systemic exposure to B17MP as Area under the concentration-time curve from zero to infinity (AUC0-∞) after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg);
Time to t1/2 of B17MPafter a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg); | From pre-dose to 24 hours post dose
  CHF 5993 BDP/FF/GB 200/6/12.5 µg pMDI vs. BDP HFA (QVAR REDIHALER®, BDP 80 µg):
  To compare the systemic exposure to B17MP as Time to t1/2 of B17MP after a single inhaled dose of CHF 5993 BDP/FF/GB 200/6/12.5 μg and of BDP HFA (QVAR REDIHALER®, BDP 80 μg);
Incidence of Adverse events | through study completion, an average of 90 days, screening phase inclusive
  Number and percentage of subject with at least one event and number of treatment-emergent events.
Incidence of study drugs reactions | through study completion, an average of 90 days, screening phase inclusive
  Number and percentage of subject with at least one event and number of treatment-emergent events.
Change of systolic and diastolic Blood pressure | from pre-dose to 24hours post dose
  The number and percentage of subjects with QTcF in the following intervals will be presented at each post-dose time point and at any post-dose time point by treatment:
  • Change from pre-dose >20 mmHg for SBP; Change from pre-dose >10 mmHg for DBP.
12-lead ECG | From Pre-dose to 75 minutes post dose
  The number and percentage of subjects with abnormal actual QTcF (Fridericia-correctedQT Interval).
12-lead ECG | From Pre-dose to 75 minutes post dose
  The number and percentage of subjects with abnormal change from the baseline of QTcF
Number of participants with abnormal laboratory test results | through study completion, an average of 90 days, screening phase inclusive
  Clinical chemistry,Fasting serum glucose;Haematology parameters will be evaluated. For continuous laboratory parameters, the laboratory values and the change from baseline will be summarised at each visit by treatment sequence using descriptive statistics. For categorical laboratory parameters, a frequency table of results will be produced at each visit by treatment sequence.
body temperature abnormal values | through study completion, an average of 90 days, screening phase inclusive
  For continuous laboratory parameters, the laboratory values and the change from baseline will be summarised at each visit by treatment sequence using descriptive statistics.
Number of participants with abnormal results of physical examinations | through study completion, an average of 90 days, screening phase inclusive
  For continuous laboratory parameters, the laboratory values and the change from baseline will be summarised at each visit by treatment sequence using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Klein, MD, Principal Investigator — SGS Belgium NV-Clinical Pharmacology Unit
Locations (1):
- SGS Belgium NV - Clinical Pharmacology Unit, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No